CLINICAL TRIAL: NCT03737955
Title: A Phase 2 Trial of Fractionated Gemtuzumab Ozogamicin to Eradicate Measurable Residual Disease in Acute Myeloid Leukemia Patients (GO for MRD)
Brief Title: Fractionated Gemtuzumab Ozogamicin in Treating Measurable Residual Disease in Patients With Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1018001; NCI-2018-01613 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9966 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2018-11-02; First posted 2018-11-13 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: Myeloid and Monocytic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Monocytic, Acute | interventions — Gemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (gemtuzumab ozogamicin) (Experimental): Patients receive gemtuzumab ozogamicin IV on days 1, 4, 7. Treatment continues for 35 days in the absence of disease progression or unacceptable toxicity. Responders and non-responders, without significant adverse events during the first course, may receive a second course of gemtuzumab ozogamicin within 60 days after course 1.
  Interventions: Drug: Gemtuzumab Ozogamicin; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Gemtuzumab Ozogamicin — Receive IV
  Other Names: CDP-771; Calicheamicin-Conjugated Humanized Anti-CD33 Monoclonal Antibody; Mylotarg
Other: Quality-of-Life Assessment — Ancillary studies

SUMMARY:
This phase II trial studies the how well fractionated gemtuzumab ozogamicin works in treating measurable residual disease in patients with acute myeloid leukemia. Gemtuzumab ozogamicin is a monoclonal antibody, called gemtuzumab, linked to a chemotherapy drug, called ozogamicin. Gemtuzumab is a form of targeted therapy because it attaches to specific molecules (receptors) on the surface of cancer cells, known as CD33 receptors, and delivers a chemotherapy known as calicheamicin to kill them.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive gemtuzumab ozogamicin intravenously (IV) on days 1, 4, 7. Treatment continues for 35 days in the absence of disease progression or unacceptable toxicity. Responders and non-responders, without significant adverse events during the first course, may receive a second course of gemtuzumab ozogamicin within 60 days after course 1.

After completion of study treatment, patients are followed up for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Prior diagnosis AML based on 2016 World Health Organization criteria. Acute promyelocytic leukemia (APL) and biphenotypic AML are not eligible
* Patients must have MRD-level disease only and otherwise meet criteria for complete response (CR) or complete remission with incomplete hematologic recovery (CRi) per the 2017 European Leukemia Net response criteria (< 5% blasts in the marrow without a requirement for peripheral blood count recovery). MRD must be measurable by multiparameter flow cytometry (MPFC) and/or polymerase chain reaction (PCR)-based molecular markers and/or karyotypic markers (e.g., classical cytogenetics or fluorescence in situ hybridization). MRD status will be centrally confirmed by the UW/FHCRC clinical laboratory in order to standardize response assessment following administration of study therapy.
* Patients must have received at least 1 cycle of standard induction chemotherapy prior to enrollment on the study. However, adult patients (>= 18 years of age) are eligible for participation at any time point in treatment (after induction, during or after consolidation, pre-transplant, or post-transplant).
* Age >= 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status =< 3
* Patient's AML blasts must have CD33 expression.
* For adults (>= 18 years of age): Serum creatinine =< 2.0 mg/dL.
* For adults (>= 18 years of age): Total bilirubin =< 2 x institutional upper limit of normal for age (unless known history of Gilbert's disease).
* For adults (>= 18 years of age): Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 x institutional upper limit of normal for age (unless thought to be related to resolving infectious complications).
* Ability of patient to provide written informed consent.
* Females of childbearing potential must have a negative pregnancy test prior to receiving GO.
* Patients who re-enroll must have achieved an MRD-negative CR during their prior enrollment

Exclusion Criteria:

* Subjects who have had chemotherapy or radiation therapy within 14 days prior to entering the study.
* Subjects may not be receiving other investigational agents.
* Uncontrolled or concurrent illness including, but not limited to, uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-11-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical response rate | Up to 70 days
  Measured by clearance of measurable residual disease (MRD) with bone marrow evaluation after one or two cycles of therapy and compare responses (rate of eradication of MRD) based on CD33 single nucleotide polymorphism rs12459419 genotype.

SECONDARY OUTCOMES:
Rate of sinusoidal obstructive syndrome (SOS) | Up to 6 months
  Measured by grade III/IV non-hematologic toxicities using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.
Rate of allogeneic hematopoietic cell transplantation (HCT) | Up to 6 Months
  Measured by those receiving HCT

CONTACTS AND LOCATIONS:
Overall Officials: Mary-Elizabeth Percival, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Center/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No